CLINICAL TRIAL: NCT06364657
Title: Role of Neurotrophic Keratitis Versus Severity of Tear Film and Ocular Surface Parameters in Determining the Differences in Corneal Structure and Function in Patients With Sjogrens vs. Non-Sjogrens Dry Eye
Brief Title: Differences in Corneal Structure and Function in Patients With Sjogrens vs. Non-Sjogrens Dry Eye
Acronym: IIR
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely closed to enrollment due to the principal investigator's departure from the institution (Johns Hopkins University).
Sponsor: Johns Hopkins University (Other)
Collaborators: Dompe U.S. Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00439625
Record Dates: First submitted 2024-04-04; First posted 2024-04-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Sjogren's Syndrome; Dry Eye; Neurotrophic Keratitis
Keywords: Sjogren's Syndrome; Dry Eye; Neurotrophic Keratitis
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sjogren's related dry-eye: Patients over the age of 18 years with known dry eye with underlying Sjogren's syndrome. Includes a previous diagnosis of dry eye made by an eye care specialist and a previous diagnosis of Sjogren's made according to the 2016 revised Sjogren's classification criteria.
  Interventions: Diagnostic Test: Eye Exam
- non-Sjogren's related dry-eye: Patients over the age of 18 years with known dry eye without underlying Sjogren's syndrome. Includes a previous diagnosis of dry eye made by an eye care specialist and a previous diagnosis of Sjogren's according to the 2016 revised Sjogren's classification criteria was definitively excluded
  Interventions: Diagnostic Test: Eye Exam
- Control: Age-matched healthy controls with no known history of ocular surface diseases or dry eye or any underlying autoimmune disease
  Interventions: Diagnostic Test: Eye Exam

INTERVENTIONS:
Diagnostic Test: Eye Exam — * Symptom Questionnaires (OSDI, eye dryness VAS, visual fatigue VAS, eye discomfort VAS)
  * Pain scale questionnaire [Wong-Baker Faces Pain Rating Scale and Ocular Pain Assessment Survey
  * Best spectacle-corrected visual acuity (BSCVA) as measured by Snellen chart followed by Mars contrast sensitivity test.
  * Corneal esthesiometer for measurement of corneal sensation
  * Schirmer's without topical anesthesia
  * Corneal epithelial thickness sand endothelial cell count using Anterior Segment Optical Coherence Tomography (AS-OCT)
  * Staining for dry eye:
  * Tear film break-up time (BUT) using fluorescein.
  * Fluorescein staining (National Eye Institute (NEI) and Ocular staining score (OSS))
  * Lissamine green staining (OSS and Oxford)
  * Non-contact confocal biomicroscopy for morphology of the ocular surface

SUMMARY:
In this study the investigators plan to enroll three groups of patients: non-Sjogren's dry eye, Sjogren's dry eye and controls. The study has the following primary goals:

1. To determine whether dry eye is associated with reduced corneal sensation
2. To determine whether reduced corneal sensation is due to the severity of the dry eye, the type of dry eye (primarily aqueous deficient versus primarily evaporative) or entirely related to the presence of Sjogren's
3. To determine whether corneal sensation is associated with ocular or systemic pain symptoms Additionally, the study aims to compare the novel corneal esthesiometer measurements to confocal biomicroscopy findings in determining neurotrophic keratitis (NK) and assess correlations between corneal sensation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older
* Capacity to give informed consent
* Self-reported literacy
* Best corrected visual acuity at distance 20/40 in each eye
* Signed Institutional Review Board (IRB)-approved consent agreeing to the terms of the study For Sjogren's-related dry eye, the below inclusion criteria will be required

  * a previous diagnosis of dry eye made by an eye care specialist
  * a previous diagnosis of Sjogren's made according to the 2016 revised Sjogren's classification criteria

Exclusion Criteria:

* ● Age less than 18 years

  * Physical or mental issues, illiteracy, or language problems that might possibly interfere with reading ability or other condition that would preclude successful participation in this study
  * Contact lens wear within 10 days of enrollment
  * Any intraocular surgery (including cataract surgery) within the last 3 months
  * Any minor ocular surgery including tear duct cauterization or plugs within the last 30 days
  * Any history of corneal surgery (including LASIK/PRK) or cosmetic lid surgery in the past 12 months
  * Any history of glaucoma surgery (e.g., trabeculectomy or a tube shunt)
  * Best corrected vision worse than 20/40
  * Known history of severe ocular surface disease that might cause corneal haze and interfere with corneal staining score including but not limited to graft-versus-host disease, mucous membrane pemphigoid, atopic keratoconjunctivitis
  * Presence of keratoconus
  * Concurrent epithelial corneal disease or dystrophy (e.g., anterior basement membrane disease, pterygium, or scarring) that might affect the corneal staining score
  * Previous use of OXERVATE® for neurotrophic keratitis
  * Neurotrophic keratoconjunctivitis or corneal/conjunctival scarring (history of herpes simplex virus or varicella zoster virus keratitis)
  * Any blepharitis eyelid procedures such as Intense Pulsed Light (IPL), low level light treatment therapy, LipiFlow®, or nasolacrimal duct probing in the last 30 days prior to the study visit
  * Any acupuncture or physical therapy on the face or head within the past 3 months
  * Current smoker (within the past year)
  * Pregnant or nursing
  * Artificial tear use within 2 hours of study visit
  * Topical ophthalmic non-steroidal anti-inflammatory drug use 24 hours before the study visit
  * History of taking or current use of topical glaucoma drops or neurostimulation drugs or devices for treating dry eye
  * History or current intravitreal injections for macular degeneration
  * History of continuous positive airway pressure usage in the past 3 months
  * Any concurrent medical condition that in the judgment of the PI might interfere with the conduct of the study, confound the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older, with and without Sjogren's-related dry eye, and no previous diagnosis of dry eye or other ocular surface disease.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Corneal Epithelium health | 1 Day
  Measuring epithelial staining score and epithelial thickness map using anterior segment Optical coherence tomography (OCT)
Corneal Nerve health | 1 Day
  Corneal sensation using non-contact esthesiometer and corneal nerve density and morphology using non-contact confocal biomicroscopy

SECONDARY OUTCOMES:
Correlations Between Corneal Staining Score | 1 Day
  Correlations between corneal staining score with visual parameters, epithelial thickness map, corneal nerve density and morphology, and corneal sensation
Correlations Between Patient Symptoms | 1 Day
  Correlations between the patient symptoms and above corneal findings using Ocular Surface Disease Index (OSDI), Visual Acuity Scale (VAS), and pain scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Esen K Akpek, MD, Principal Investigator — Johns Hopkins Hospital Wilmer Eye Institute
Locations (1):
- Johns Hopkins Hospital Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No